CLINICAL TRIAL: NCT06655701
Title: Stress Urinary Incontinence and Sarcopenia in Postmenopausal Osteoporosis: The Intersection of Muscle Loss and Pelvic Dysfunction
Brief Title: Stress Urinary Incontinence and Sarcopenia in Postmenopausal Osteoporosis
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH8
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal osteoporosis: Postmenopausal osteoporosis is diagnosed using Dual-X-ray Absorptiometry (DXA), which measures bone mineral density (BMD) and provides a T-score. A T-score of -2.5 or lower confirms the diagnosis of osteoporosis.
  Interventions: Diagnostic Test: No intervention
- Postmenopausal non-osteoporotic women: These women maintain normal bone mineral density (BMD) levels, typically assessed using Dual-X-ray Absorptiometry (DXA). A T-score above -1.0 is considered normal.
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
The primary aim of our study is to evaluate the presence of stress urinary incontinence in postmenopausal patients with and without osteoporosis, determine its impact on quality of life, and explore its relationship with sarcopenia.

DETAILED DESCRIPTION:
One hundred postmenopausal women, aged 50-75, who applied to the Physical Therapy and Rehabilitation outpatient clinic at Beylikdüzü State Hospital and have Dual-X-ray Absorptiometry (DXA) measurements taken within the last 6 months, including both osteoporotic and non-osteoporotic patients, will be included in the study. Sociodemographic data such as age, gender, height, weight, and BMI will be recorded. DXA results, including femoral neck and L1-L4 T-scores and BMD values, will be obtained. Patients will be asked about osteoporosis treatment, presence of fecal incontinence, constipation, and medication use. Stress urinary incontinence will be determined through a questionnaire, and its impact on quality of life will be assessed using the Incontinence Quality of Life Scale. In the second phase, sarcopenia will be evaluated according to the Asian Working Group for Sarcopenia (AWGS) criteria by assessing skeletal muscle mass (via bioelectrical impedance analysis), handgrip strength, and the 5-times sit-to-stand test.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with DXA measurements performed within the last 6 months.
* Based on DXA measurements:

Femoral neck and L1-L4 T-scores of -1 and above will be included in the control group (non-osteoporotic).

Femoral neck and L1-L4 T-scores of -2.5 and below will be included in the osteoporosis group.

* Aged 50-75 years

Exclusion Criteria:

* Refusal to participate in the study.
* History of neurological diseases, infections, surgeries, or trauma that could cause urinary incontinence or muscle loss.
* Presence of psychiatric disorders.
* Cognitive impairments.
* Use of medications that could affect the study results.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Presence of Stress Urinary Incontinence: | 0 day
  Stress urinary incontinence (SUI) is the involuntary leakage of urine during physical activities that increase abdominal pressure, such as coughing, sneezing, or lifting. In this study, the presence of SUI will be determined through a questionnaire that asks participants about symptoms and frequency of urine leakage during such activities.
Incontinence Quality of Life Scale (I-QOL): | 0 day
  The I-QOL is a validated questionnaire that measures the impact of urinary incontinence on a patient's quality of life. It assesses how incontinence affects daily activities, social interactions, and emotional well-being. Higher scores indicate better quality of life, while lower scores suggest that incontinence has a more significant negative impact on the patient's day-to-day functioning.
Skeletal Muscle Mass: | 0 day
  Measured by bioelectrical impedance analysis (BIA), this assesses the amount of muscle tissue in the body. Low skeletal muscle mass indicates sarcopenia.
Handgrip Strength | 0 day
  This is a simple test to measure muscle strength. Reduced handgrip strength is a sign of sarcopenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No